CLINICAL TRIAL: NCT00421148
Title: A Multi-Center, Randomized, Parallel Dose-Finding, Safety Assessor-Blinded Trial to Explore the Efficacy, Safety and Pharmacokinetics of Four Doses of Org 25969 and Placebo in Pediatric and Adult Subjects.
Brief Title: Dose-Finding Pediatric and Adult Trial With Sugammadex (Org 25969, MK-8616, SCH 900616) (19.4.306) (MK-8616-034) (P05961)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05961; 2004-003819-23 (EudraCT Number); 19.4.306 (Other: Organon Protocol Number); MK-8616-034 (Other: Merck Protocol Number); P05961 (Other: Schering-Plough Protocol Number)
Record Dates: First submitted 2007-01-08; First posted 2007-01-11 (Estimated); Results first posted 2019-01-28 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2018-08

CONDITIONS: Anesthesia
MeSH Terms: interventions — Sugammadex; Sodium Chloride; Solutions; Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Sugammadex 0.5 mg/kg (Experimental): Participants are to receive an intravenous (IV) single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single bolus dose of 0.5 mg/kg sugammadex is to be given.
  Interventions: Drug: Sugammadex 0.5 mg/kg; Drug: Rocuronium bromide
- Sugammadex 1 mg/kg (Experimental): Participants are to receive an IV single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single bolus dose of 1 mg/kg sugammadex is to be given.
  Interventions: Drug: Sugammadex 1 mg/kg; Drug: Rocuronium bromide
- Sugammadex 2 mg/kg (Experimental): Participants are to receive an IV single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single bolus dose of 2 mg/kg sugammadex is to be given.
  Interventions: Drug: Sugammadex 2 mg/kg; Drug: Rocuronium bromide
- Sugammadex 4 mg/kg (Experimental): Participants are to receive an IV single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single bolus dose of 4 mg/kg sugammadex is to be given.
  Interventions: Drug: Sugammadex 4 mg/kg; Drug: Rocuronium bromide
- Placebo (Placebo Comparator): Participants are to receive an IV single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single 3-mL bolus dose of placebo (sodium chloride 0.9% solution) is to be given.
  Interventions: Drug: Placebo; Drug: Rocuronium bromide

INTERVENTIONS:
Drug: Sugammadex 0.5 mg/kg — IV infusion
  Other Names: Org 25969; MK-8616; SCH 900616
  Arms: Sugammadex 0.5 mg/kg
Drug: Sugammadex 1 mg/kg — IV infusion
  Other Names: Org 25969; MK-8616; SCH 900616
  Arms: Sugammadex 1 mg/kg
Drug: Sugammadex 2 mg/kg — IV infusion
  Other Names: Org 25969; MK-8616; SCH 900616
  Arms: Sugammadex 2 mg/kg
Drug: Sugammadex 4 mg/kg — IV infusion
  Other Names: Org 25969; MK-8616; SCH 900616
  Arms: Sugammadex 4 mg/kg
Drug: Placebo — IV infusion
  Other Names: sodium chloride 0.9% solution
  Arms: Placebo
Drug: Rocuronium bromide — IV infusion
  Other Names: ESMERON®

SUMMARY:
The purpose of this study is:

* to explore the dose-response relation of sugammadex (Org 25969, MK-8616, SCH 900616) given as a reversal agent at reappearance of T2 after 0.6 mg.kg-1 rocuronium in pediatric and adult participants
* to explore the pharmacokinetics (PK) of sugammadex in pediatric and adult participants, and to evaluate the safety of sugammadex in pediatric and adult participants.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class 1 - 2, between the ages of 28 days and 65 years inclusive, and between the ages of 2 and 65 years inclusive for Germany and between the ages of 6 and 65 years inclusive for Finland
* Scheduled for general anesthesia with an anticipated duration of anesthesia of at least 60 minutes, without further need for muscle relaxation other than one single dose of 0.6 mg/kg rocuronium
* Scheduled for surgical procedures in the supine position
* Participants who, and/or whose parent(s) or legal guardian(s) have given written informed consent [or appropriate assent, if applicable]

Exclusion Criteria:

* Known or suspected neuromuscular disorders impairing neuromuscular blockade (NMB) and/or significant renal dysfunction, in Germany creatinine and blood urea nitrogen outside local reference ranges
* Known or suspected to have a (family) history of malignant hyperthermia
* Known or suspected to have an allergy to narcotics, muscle relaxants or other medication used during general anesthesia
* Use of medication expected to interfere with the rocuronium given in this trial, based on the dose and the time of administration
* Pregnancy
* Childbearing potential not using any of the following methods of birth control: condom or diaphragm with spermicide, vasectomized partner (>6 months), intrauterine device (IUD), abstinence
* Breast-feeding
* Prior participation in any study with Org 25969 (sugammadex)
* Participation in another clinical trial, not pre-approved by NV Organon, within 30 days of entering into study 19.4.306 (MK-8616-034, P05961)

Ages: 28 Days to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2005-05-30 (Actual); Primary Completion 2006-05-31 (Actual); Study Completion 2006-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Plaud B, Meretoja O, Hofmockel R, Raft J, Stoddart PA, van Kuijk JH, Hermens Y, Mirakhur RK. Reversal of rocuronium-induced neuromuscular blockade with sugammadex in pediatric and adult surgical patients. Anesthesiology. 2009 Feb;110(2):284-94. doi: 10.1097/ALN.0b013e318194caaa. PMID 19194156
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited participants were stratified between Infants (28 days-23 months of age), Children (2-11 years of age), Adolescents (12-17 years of age) and Adults (18-65 years of age). For Participant Flow, participants are included in the treatment group to which they were randomized.
Pre-assignment Details: One adolescent participant was inadvertently randomized to Children: Sugammadex 4 mg/kg, but was included in Adolescents: Sugammadex 4 mg/kg for safety analyses. One participant was randomized to Adolescents: Sugammadex 0.5 mg/kg, but received sugammadex 5.0 mg/kg & was included in the Adolescents: Sugammadex 4 mg/kg for safety analyses.
Groups:
- Infants: Placebo: Infant participants received an intravenous (IV) single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single bolus dose of placebo (sodium chloride 0.9% solution) was administered.
- Infants: Sugammadex 0.5 mg/kg: Infant participants received an IV single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single bolus dose of 0.5 mg/kg sugammadex was administered.
- Infants: Sugammadex 1 mg/kg: Infant participants received an IV single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single bolus dose of 1 mg/kg sugammadex was administered.
- Infants: Sugammadex 2 mg/kg: Infant participants received an IV single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single bolus dose of 2 mg/kg sugammadex was administered.
- Infants: Sugammadex 4 mg/kg: Infant participants received an IV single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single bolus dose of 4 mg/kg sugammadex was administered.
- Children: Placebo: Child participants received an IV single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single bolus dose of placebo (sodium chloride 0.9% solution) was administered.
- Children: Sugammadex 0.5 mg/kg: Child participants received an IV single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single bolus dose of 0.5 mg/kg sugammadex was administered.
- Children: Sugammadex 1 mg/kg: Child participants received an IV single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single bolus dose of 1 mg/kg sugammadex was administered
- Children: Sugammadex 2 mg/kg: Child participants received an IV single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single bolus dose of 2 mg/kg sugammadex was administered.
- Children: Sugammadex 4 mg/kg: Child participants received an IV single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single bolus dose of 4 mg/kg sugammadex was administered.
- Adolescents: Placebo: Adolescent participants received an IV single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single bolus dose of placebo (sodium chloride 0.9% solution) was administered.
- Adolescents: Sugammadex 0.5 mg/kg: Adolescent participants received an IV single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single bolus dose of 0.5 mg/kg sugammadex was administered.
- Adolescents: Sugammadex 1 mg/kg: Adolescents participants received an IV single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single bolus dose of 1 mg/kg sugammadex was administered.
- Adolescents: Sugammadex 2 mg/kg: Adolescent participants received an IV single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single bolus dose of 2 mg/kg sugammadex was administered.
- Adolescents: Sugammadex 4 mg/kg: Adolescent participants received an IV single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single bolus dose of 4 mg/kg sugammadex was administered.
- Adults: Placebo: Adult participants received an IV single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single bolus dose of placebo (sodium chloride 0.9% solution) was administered.
- Adults: Sugammadex 0.5 mg/kg: Adult participants received an IV single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single bolus dose of 0.5 mg/kg sugammadex was administered.
- Adults: Sugammadex 1 mg/kg: Adult participants received an IV single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single bolus dose of 1 mg/kg sugammadex was administered.
- Adults: Sugammadex 2 mg/kg: Adult participants received an IV single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single bolus dose of 2 mg/kg sugammadex was administered.
- Adults: Sugammadex 4 mg/kg: Adult participants received an IV single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single bolus dose of 4 mg/kg sugammadex was administered.
Period: Overall Study
Arm/Group | Infants: Placebo | Infants: Sugammadex 0.5 mg/kg | Infants: Sugammadex 1 mg/kg | Infants: Sugammadex 2 mg/kg | Infants: Sugammadex 4 mg/kg | Children: Placebo | Children: Sugammadex 0.5 mg/kg | Children: Sugammadex 1 mg/kg | Children: Sugammadex 2 mg/kg | Children: Sugammadex 4 mg/kg | Adolescents: Placebo | Adolescents: Sugammadex 0.5 mg/kg | Adolescents: Sugammadex 1 mg/kg | Adolescents: Sugammadex 2 mg/kg | Adolescents: Sugammadex 4 mg/kg | Adults: Placebo | Adults: Sugammadex 0.5 mg/kg | Adults: Sugammadex 1 mg/kg | Adults: Sugammadex 2 mg/kg | Adults: Sugammadex 4 mg/kg
Started | 2 | 2 | 2 | 1 | 1 | 5 | 6 | 5 | 5 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Treated | 2 | 2 | 2 | 1 | 1 | 4 (1 additional participant discontinued prior to receiving study treatment) | 6 | 5 | 5 | 5 (Includes 1 participant who was inadvertently randomized to group but was an adolescent) | 6 | 6 (Includes 1 participant who was inadvertently randomized to group but received 5 mg/kg sugammadex) | 6 | 6 | 6 | 6 | 6 | 5 (1 additional participant discontinued prior to receiving study treatment) | 5 (1 additional participant discontinued prior to receiving study treatment) | 6
Completed | 2 | 2 | 2 | 1 | 1 | 4 | 6 | 5 | 5 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The All-Participants-Treated (APT) population consisted of all treated participants. Three additional participants withdrew from the study before receiving treatment & were not included in the Baseline Analysis Population. For the APT population, participants with incorrect randomization are included under the actual dose group they received.
Groups:
- Infants: Placebo: Infant participants received an IV single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single bolus dose of placebo (sodium chloride 0.9% solution) was administered.
- Total: Total of all reporting groups
Arm/Group | Infants: Placebo | Infants: Sugammadex 0.5 mg/kg | Infants: Sugammadex 1 mg/kg | Infants: Sugammadex 2 mg/kg | Children: Placebo | Children: Sugammadex 0.5 mg/kg | Children: Sugammadex 1 mg/kg | Children: Sugammadex 2 mg/kg | Children: Sugammadex 4 mg/kg | Adolescents: Placebo | Adolescents: Sugammadex 0.5 mg/kg | Adolescents: Sugammadex 1 mg/kg | Adolescents: Sugammadex 2 mg/kg | Adolescents: Sugammadex 4 mg/kg | Adults: Placebo | Adults: Sugammadex 0.5 mg/kg | Adults: Sugammadex 1 mg/kg | Adults: Sugammadex 2 mg/kg | Adults: Sugammadex 4 mg/kg | Infants: Sugammadex 4 mg/kg | Total
Number analyzed (Participants) | 2 | 2 | 2 | 1 | 4 | 6 | 5 | 5 | 4 | 6 | 5 | 6 | 6 | 8 | 6 | 6 | 5 | 5 | 6 | 1 | 91
Age, Continuous [Mean (Standard Deviation); unit: Years] | 1 (0) | 1 (0) | 1 (0) | 0 (NA) — NA=Not calculated on 1 participant | 9 (1) | 9 (3) | 8 (2) | 9 (2) | 6 (3) | 15 (2) | 14 (1) | 15 (2) | 14 (0) | 14 (2) | 49 (12) | 41 (17) | 37 (8) | 38 (10) | 38 (14) | 1 (NA) — NA=Not calculated on 1 participant | 19.8 (16.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 0 | 1 | 5 | 3 | 3 | 2 | 3 | 0 | 3 | 3 | 4 | 0 | 2 | 2 | 1 | 2 | 0 | 38
  Male | 0 | 0 | 2 | 1 | 3 | 1 | 2 | 2 | 2 | 3 | 5 | 3 | 3 | 4 | 6 | 4 | 3 | 4 | 4 | 1 | 53

OUTCOME MEASURES:

1. Primary Outcome: Time From Start of Administration of Study Treatment (Sugammadex or Placebo) to Recovery T4/T1 Ratio to 0.9
Description: Neuromuscular functioning was monitored by applying repetitive Train-Of-Four (TOF) electrical stimulations to the ulnar nerve every 15 seconds & assessing twitch response at the adductor pollicis muscle. T1 & T4 refer to the magnitudes (heights) of the first & fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from neuromuscular blockade (NMB). In this study, twitch responses were recorded until the T4/T1 Ratio reached ≥0.9, the minimum acceptable ratio that indicated recovery from NMB. A faster time to recovery of the T4/T1 Ratio to 0.9 indicates a faster recovery from NMB.
Time Frame: From start of sugammadex or palcebo administration to recovery of T4/T1 ratio to 0.9 (ranging from ~0.5 minutes to ~30 minutes from sugammadex or placebo administration)
Population: The Per Protocol (PP) population consisted of all randomized participants who received a dose of study treatment (sugammadex or placebo) & had ≥1 post-baseline efficacy measurement for this outcome measure & had no protocol violations. For efficacy, participants with incorrect randomization were included under the planned dose group.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Infants: Placebo | Infants: Sugammadex 0.5 mg/kg | Infants: Sugammadex 1 mg/kg | Infants: Sugammadex 2 mg/kg | Children: Placebo | Children: Sugammadex 0.5 mg/kg | Children: Sugammadex 1 mg/kg | Children: Sugammadex 2 mg/kg | Children: Sugammadex 4 mg/kg | Adolescents: Placebo | Adolescents: Sugammadex 0.5 mg/kg | Adolescents: Sugammadex 1 mg/kg | Adolescents: Sugammadex 2 mg/kg | Adolescents: Sugammadex 4 mg/kg | Adults: Placebo | Adults: Sugammadex 0.5 mg/kg | Adults: Sugammadex 1 mg/kg | Adults: Sugammadex 2 mg/kg | Adults: Sugammadex 4 mg/kg | Infants: Sugammadex 4 mg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 1 | 4 | 5 | 5 | 4 | 4 | 5 | 5 | 6 | 6 | 6 | 6 | 5 | 5 | 5 | 5 | 1
Minutes | 20.98 (11.30) | 3.72 (0.63) | 2.42 (0.70) | 0.58 (NA) — NA=Not calculated on 1 participant | 19.57 (10.97) | 5.22 (3.50) | 3.95 (3.23) | 1.20 (0.35) | 1.57 (1.90) | 22.77 (13.10) | 11.97 (17.65) | 1.77 (0.37) | 1.87 (1.70) | 1.08 (0.25) | 29.48 (8.43) | 3.77 (1.12) | 1.62 (0.30) | 1.27 (0.27) | 1.37 (0.38) | 0.67 (NA) — NA=Not calculated on 1 participant

2. Secondary Outcome: Time From Start of Administration of Study Treatment (Sugammadex or Placebo) to Recovery T4/T1 Ratio to 0.7
Description: Neuromuscular functioning was monitored by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds & assessing twitch response at the adductor pollicis muscle. T1 & T4 refer to the magnitudes (heights) of the first & fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from NMB. A faster time to recovery of the T4/T1 Ratio to 0.7 indicates a faster recovery from NMB.
Time Frame: From start of sugammadex or placebo administration to recovery of T4/T1 ratio to 0.7 (ranging from ~0.4 minutes to ~20 minutes from sugammadex or placebo administration)
Population: The PP population consisted of all randomized participants who received a dose of study treatment (sugammadex or placebo) & had ≥1 post-baseline efficacy measurement for this outcome measure & had no protocol violations. For efficacy, participants with incorrect randomization were included under the planned dose group.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Infants: Placebo | Infants: Sugammadex 0.5 mg/kg | Infants: Sugammadex 1 mg/kg | Infants: Sugammadex 2 mg/kg | Children: Placebo | Children: Sugammadex 0.5 mg/kg | Children: Sugammadex 1 mg/kg | Children: Sugammadex 2 mg/kg | Children: Sugammadex 4 mg/kg | Adolescents: Placebo | Adolescents: Sugammadex 0.5 mg/kg | Adolescents: Sugammadex 1 mg/kg | Adolescents: Sugammadex 2 mg/kg | Adolescents: Sugammadex 4 mg/kg | Adults: Placebo | Adults: Sugammadex 0.5 mg/kg | Adults: Sugammadex 1 mg/kg | Adults: Sugammadex 2 mg/kg | Adults: Sugammadex 4 mg/kg | Infants: Sugammadex 4 mg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 1 | 4 | 5 | 5 | 4 | 4 | 6 | 5 | 6 | 6 | 6 | 6 | 5 | 5 | 5 | 5 | 1
Minutes | 14.85 (8.65) | 2.47 (0.07) | 1.78 (0.18) | 0.58 (NA) — NA=Not calculated on 1 participant | 12.32 (7.00) | 2.62 (0.93) | 1.45 (0.38) | 0.75 (0.12) | 0.57 (0.13) | 18.62 (9.72) | 2.77 (1.27) | 1.07 (0.12) | 0.95 (0.30) | 0.83 (0.20) | 19.65 (5.38) | 1.62 (0.25) | 1.27 (0.35) | 0.87 (0.23) | 1.12 (0.38) | 0.42 (NA) — NA=Not calculated on 1 participant

3. Secondary Outcome: Time From Start of Administration of Study Treatment (Sugammadex or Placebo) to Recovery T4/T1 Ratio to 0.8
Description: Neuromuscular functioning was monitored by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds & assessing twitch response at the adductor pollicis muscle. T1 & T4 refer to the magnitudes (heights) of the first & fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from NMB. A faster time to recovery of the T4/T1 Ratio to 0.8 indicates a faster recovery from NMB.
Time Frame: From start of sugammadex or placebo administration to recovery of T4/T1 ratio to 0.8 (ranging from ~0.5 minutes to ~25 minutes from sugammadex or placebo administration)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Infants: Placebo | Infants: Sugammadex 0.5 mg/kg | Infants: Sugammadex 1 mg/kg | Infants: Sugammadex 2 mg/kg | Children: Placebo | Children: Sugammadex 0.5 mg/kg | Children: Sugammadex 1 mg/kg | Children: Sugammadex 2 mg/kg | Children: Sugammadex 4 mg/kg | Adolescents: Placebo | Adolescents: Sugammadex 0.5 mg/kg | Adolescents: Sugammadex 1 mg/kg | Adolescents: Sugammadex 2 mg/kg | Adolescents: Sugammadex 4 mg/kg | Adults: Placebo | Adults: Sugammadex 0.5 mg/kg | Adults: Sugammadex 1 mg/kg | Adults: Sugammadex 2 mg/kg | Adults: Sugammadex 4 mg/kg | Infants: Sugammadex 4 mg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 1 | 4 | 5 | 5 | 4 | 4 | 6 | 5 | 6 | 6 | 6 | 6 | 5 | 5 | 5 | 5 | 1
Minutes | 17.85 (10.42) | 2.97 (0.07) | 2.03 (0.17) | 0.58 (NA) — NA=Not calculated on 1 participant | 14.20 (8.32) | 3.42 (1.40) | 1.85 (0.70) | 0.95 (0.23) | 0.75 (0.45) | 21.92 (12.52) | 4.92 (4.08) | 1.35 (0.17) | 0.98 (0.38) | 0.87 (0.18) | 24.77 (9.33) | 2.22 (0.60) | 1.37 (0.35) | 1.07 (0.23) | 1.27 (0.30) | 0.67 (NA) — NA=Not calculated on 1 participant

ADVERSE EVENTS:
Time Frame: Through postoperative Day 7 (Up to 8 days)
Description: The APT population consisted of all randomized participants who received a dose of study treatment (sugammadex or placebo). With respect to the APT population, participants with incorrect randomization were included under the actual dose group they received.
Groups:
- Infants: Sugammadex .0.5 mg/kg: Infant participants received an IV single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single bolus dose of 0.5 mg/kg sugammadex was administered.
- Adolescents: Sugammadex 1 mg/kg: Adolescent participants received an IV single bolus dose of 0.6 mg/kg rocuronium. At reappearance of T2, an IV single bolus dose of 1 mg/kg sugammadex was administered.
Arm/Group | Infants: Placebo | Infants: Sugammadex .0.5 mg/kg | Infants: Sugammadex 1 mg/kg | Infants: Sugammadex 2 mg/kg | Infants: Sugammadex 4 mg/kg | Children: Placebo | Children: Sugammadex 0.5 mg/kg | Children: Sugammadex 1 mg/kg | Children: Sugammadex 2 mg/kg | Children: Sugammadex 4 mg/kg | Adolescents: Placebo | Adolescents: Sugammadex 0.5 mg/kg | Adolescents: Sugammadex 1 mg/kg | Adolescents: Sugammadex 2 mg/kg | Adolescents: Sugammadex 4 mg/kg | Adults: Placebo | Adults: Sugammadex 0.5 mg/kg | Adults: Sugammadex 1 mg/kg | Adults: Sugammadex 2 mg/kg | Adults: Sugammadex 4 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/1 | 0/1 | 0/4 | 0/6 | 0/5 | 0/5 | 0/4 | 0/6 | 0/5 | 0/6 | 0/6 | 0/8 | 0/6 | 0/6 | 0/5 | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/2 | 0/2 | 0/1 | 0/1 | 0/4 | 0/6 | 0/5 | 0/5 | 1/4 | 0/6 | 0/5 | 0/6 | 0/6 | 0/8 | 0/6 | 0/6 | 0/5 | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 2/2 | 1/2 | 1/2 | 1/1 | 1/1 | 3/4 | 4/6 | 2/5 | 2/5 | 4/4 | 5/6 | 3/5 | 3/6 | 5/6 | 5/8 | 3/6 | 1/6 | 5/5 | 4/5 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infants: Placebo (N=2) | Infants: Sugammadex .0.5 mg/kg (N=2) | Infants: Sugammadex 1 mg/kg (N=2) | Infants: Sugammadex 2 mg/kg (N=1) | Infants: Sugammadex 4 mg/kg (N=1) | Children: Placebo (N=4) | Children: Sugammadex 0.5 mg/kg (N=6) | Children: Sugammadex 1 mg/kg (N=5) | Children: Sugammadex 2 mg/kg (N=5) | Children: Sugammadex 4 mg/kg (N=4) | Adolescents: Placebo (N=6) | Adolescents: Sugammadex 0.5 mg/kg (N=5) | Adolescents: Sugammadex 1 mg/kg (N=6) | Adolescents: Sugammadex 2 mg/kg (N=6) | Adolescents: Sugammadex 4 mg/kg (N=8) | Adults: Placebo (N=6) | Adults: Sugammadex 0.5 mg/kg (N=6) | Adults: Sugammadex 1 mg/kg (N=5) | Adults: Sugammadex 2 mg/kg (N=5) | Adults: Sugammadex 4 mg/kg (N=6)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infants: Placebo (N=2) | Infants: Sugammadex .0.5 mg/kg (N=2) | Infants: Sugammadex 1 mg/kg (N=2) | Infants: Sugammadex 2 mg/kg (N=1) | Infants: Sugammadex 4 mg/kg (N=1) | Children: Placebo (N=4) | Children: Sugammadex 0.5 mg/kg (N=6) | Children: Sugammadex 1 mg/kg (N=5) | Children: Sugammadex 2 mg/kg (N=5) | Children: Sugammadex 4 mg/kg (N=4) | Adolescents: Placebo (N=6) | Adolescents: Sugammadex 0.5 mg/kg (N=5) | Adolescents: Sugammadex 1 mg/kg (N=6) | Adolescents: Sugammadex 2 mg/kg (N=6) | Adolescents: Sugammadex 4 mg/kg (N=8) | Adults: Placebo (N=6) | Adults: Sugammadex 0.5 mg/kg (N=6) | Adults: Sugammadex 1 mg/kg (N=5) | Adults: Sugammadex 2 mg/kg (N=5) | Adults: Sugammadex 4 mg/kg (N=6)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (4) | 2 (6) | 1 (1) | 3 (3) | 3 (4) | 0 (0) | 1 (1) | 3 (4) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria traumatic (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative fever (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (2) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 3 (3) | 4 (5) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Excitability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Organon recognizes the right of the investigator(s) to publish, but all publications must be based on data validated by Organon. Any such scientific paper, presentation, or other communication concerning the clinical trial described in this protocol will first be submitted to Organon, at least six weeks ahead of estimated publication or presentation, for written consent, which shall not be withheld unreasonably.